CLINICAL TRIAL: NCT03711461
Title: Comparisons of the Risks of Gastric Distension and Delayed Recovery of Cough Reflex and Oral Intake on Intubated and Non-intubated VATS Patients
Brief Title: Recovery Between NIVATS and Intubated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201804093RIND
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Function in Thoracoscopy

STUDY DESIGN:
Intervention Model Description: intubated and nonintubated patients
Who Masked: Outcomes Assessor
Masking Description: the swallowing function assessor is blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nonintubated (Active Comparator): patients received nonintubated during thoracoscopy
  Interventions: Device: nonintubated
- intubated (Experimental): patients receiving intubated during thoracoscopy
  Interventions: Device: endotracheal tube (double lumen)

INTERVENTIONS:
Device: endotracheal tube (double lumen) — patients routinely use double lumen endotracheal intubation while they have received thoracoscopy
  Arms: intubated
Device: nonintubated — patients receiving nonintubated anesthetic plan while they have received thoracoscopy
  Arms: nonintubated

SUMMARY:
the investigator aimed to observe the changes and difference of pharyngeal function parameters between the patients receiving the intubated or nonintubated thoracoscopy by esophageal manometry, impedance, and ultrasonography

DETAILED DESCRIPTION:
Background: Anesthetic agents alter pharyngeal function with risk of impaired airway protection and aspiration. The pharyngeal function change including the swallowing and gastric regurgitation between intubated and nonintubated thoracoscopy still remains unclear.

The esophageal manometry has pressure sensor to measure the upper esophageal sphincter (UES) pressure. The manometry and impedance could detect the esophageal swallowing function during the perioperative period. The ultrasonography was used to measure the oropharyngeal swallowing function.

Objectives:the investigator aimed to observe the changes and difference of pharyngeal function parameters between the patients receiving the intubated or nonintubated thoracoscopy by esophageal manometry, impedance, and ultrasonography.

Patients and methods: Consecutive patients who will fulfill the criteria of nonintubated patients under general anesthesia and age from 20 to 80 years old will be enrolled. All subjects would receive the swallowing function by ultrasonography before the surgeries. The cough test and gastric volume were also measured. The patient was randomized by the intubated or nonintubated thoracoscopy. After induction, the endotracheal tube (ETT) will be inserted to establish airway. The non-intubated group will be use the oxygen mask and the nasal airway to maintain the airway patent. After the patients were sedated, investigators would use the video-assisted laryngoscope to let the manometry and impedance transnasal into the esophagus.These esophageal function was measured during the whole perioperative periods, especially the recovery from anesthesia in the postoperative anesthesia unit (PACU). The patients will be followed for the swallowing function by ultrasonography and cough test in the PACU, too. The oxidative test would be performed by blood test on the time, which were after anesthesia, one-lung ventilation 15 to 30 minutes, and two-lung ventilation 15 to 20 minutes, respectively.

Expected result: investigators will observe the changes between the patients receiving intubated or nonintubated thoracoscopies of the changes between the preoperative and postoperative changes in the swallowing function, cough and gastric regurgitation. The oxidative test will also be tested accompanied by the anesthetic monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfill the criteria of nonintubated thoracoscopy under general anesthesia, including tumours smaller than 6 cm, peripheral lesions, no evidence of severe adhesion; and no evidence of chest wall, diaphragm, or main bronchus involvement. Patients who had potential or confirmed airway complications such as bronchial tumor or hemothorax, morbid obesity (BMI greater than 35 kg·m-2), coagulopathy, anatomical deformity or an American Society of Anesthesiology (ASA) classification greater than 3 were excluded
2. Aged from 20-80 years old

Exclusion Criteria:

1. Major systemic disease, such as congestive heart failure, liver cirrhosis, and end stage renal disease.
2. Patients who have the risk of difficult ventilation or intubation.
3. pregnant women
4. coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-10-25 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
impedance changes | average 4 hours
  using esophageal manometry to evaluate the swallowing

SECONDARY OUTCOMES:
esophageal pressure changes | average 4 hours
  using esophageal manometry to evaluate the swallowing
hyoid bone distance | average 4 hours
  using ultrasound to evaluate the swallowing

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Ya-Jung Cheng, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided